CLINICAL TRIAL: NCT01452321
Title: Repetitive Transcranial Magnetic Stimulation Effects on Clinical, Cognitive and Social Performance in Postpartum Depression
Brief Title: Repetitive Transcranial Magnetic Stimulation in Postpartum Depression
Acronym: rTMSPPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Eduardo Moacyr Krieger, Associate Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0588/07
Record Dates: First submitted 2010-11-22; First posted 2011-10-14 (Estimated); Last update posted 2011-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Depression, Postpartum
Keywords: Transcranial Magnetic Stimulation;; Postpartum Depression;; Clinical Performance;; Cognitive Performance;; Social Performance
MeSH Terms: conditions — Depression, Postpartum | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham rTMS (Placebo Comparator): Drug-free patients, receiving 20 sessions (1 session daily) of sham (placebo) rTMS delivered to the left dorsolateral prefrontal cortex.
  Interventions: Procedure: repetitive transcranial magnetic stimulation (rTMS)
- Active rTMS (Active Comparator): Drug-free patients, receiving 20 sessions (1 session daily) of active rTMS delivered to the left dorsolateral prefrontal cortex.
  Interventions: Procedure: repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Procedure: repetitive transcranial magnetic stimulation (rTMS) — 20 daily sessions: each with 25 trains of 10 seconds at 5Hz, with a 20 second inter-train interval, at an intensity of 120% of motor threshold.
  Site: Left Dorsolateral Prefrontal Cortex
  Other Names: TMS

SUMMARY:
Several factors characterize repetitive transcranial magnetic stimulation (rTMS) as a strategic aid in the treatment of postpartum depression.

However, up to current days there have been no studies evaluating the effects of rTMS on neurocognitive and social performance of women suffering from the disorder.

The present study evaluates the impacts of rTMS in clinical, cognitive and social performance.

DETAILED DESCRIPTION:
Transcranial magnetic stimulation is a noninvasive technique that can influence specific areas of the brain and has very few side effects.

The treatment with transcranial magnetic stimulation requires attendance to hospital daily sessions for 4 consecutive weeks. Each session lasts up to 30 minutes.

Side effects include scalp discomfort and mild headache. No anesthesia is required.

Stimulation aims the dorsolateral prefrontal cortex, a region previously studied to treat depression symptoms with positive results.

The present technique has never been employed in previous studies, but risks are insignificant.

ELIGIBILITY:
Inclusion Criteria:

* major depression with a puerperal onset, according to the criteria of the DSM-IV-R (APA, 2000), as well as through a structured clinical interview (SCID-1/P v 2.0)
* baseline score of at least 14 points on the Hamilton Depression rating Scale-17 items
* baseline score of at least 13 points on the Edinburgh Postnatal Depression Scale.
* range = 18-36 years
* women who had given birth 1-6 months
* any pharmacological treatment other than clonazepam (1 mg/day)

Exclusion Criteria:

* comprised ferromagnetic metallic implants
* pacemakers
* previous neurosurgery
* history of seizures
* major head trauma
* alcoholism
* drug addiction
* any psychiatric or neurological disorder other than depression and anxiety
* psychotic depression
* suicidal propensities

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS) | 6 weeks
  Reduction on the scores of HDRS (as on the scores of Edinburgh Pospartum Depression Scale and Hamilton Anxiety Scale; and improves the global clinical status in Clinical Global Impression, Global Assessment Scale and 36-item Short-form Health Survey - Quality of Life)

SECONDARY OUTCOMES:
Battery of Neuropsychological Tests and Social Adjustment Scale | 6 weeks
  Performance of neuropsychological tests and social function - Trail Making Test, Wisconsin Card Sorting Test, Controlled Oral Word Association Test, Victoria Stroop Test, Rey Auditory Verbal Learning Test, WAIS-III (adapted for use in Brazil) subtests Similarities, Picture Completion, Digit Span, Digit-Symbol Coding and Social Adjustment Scale-Self Report (SAS-SR; adapted for use in Brazil)

CONTACTS AND LOCATIONS:
Overall Officials: Martin L Myczkowski, MSD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Department and Institute of Psychiatry, General Hospital, University of Sao Paulo medical school, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Garcia KS, Flynn P, Pierce KJ, Caudle M. Repetitive transcranial magnetic stimulation treats postpartum depression. Brain Stimul. 2010 Jan;3(1):36-41. doi: 10.1016/j.brs.2009.06.001. Epub 2009 Jul 8. PMID 20633429